CLINICAL TRIAL: NCT05696054
Title: Diagnostic Performance of Different Scores for Predicting Spontaneous Bacterial Peritonitis in Cirrhotic Patients
Brief Title: Laboratory Diagnosis of Spontaneous Bacterial Peritonitis
Acronym: SBP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Maher, Lecturer of Tropical Medicine and Gastroenterology, Sohag University
Other Study IDs: 246810
Record Dates: First submitted 2023-01-01; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample Ascitic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBP group: Patients diagnosed as spontaneous bacterial peritonitis based on ascitic fluid study.
- non-SBP group: Patients without spontaneous bacterial peritonitis based on ascitic fluid study

SUMMARY:
This study aims at evaluating the diagnostic accuracy of serum procalcitonin, PEC index, modified Wehmeyer, and Mansoura scoring systems for SBP in cirrhotic patients with ascites

DETAILED DESCRIPTION:
Based on clinical diagnosis, SBP is commonly underdiagnosed because of its nonspecific or asymptomatic presentation. Therefore, a diagnostic paracentesis should be performed in all cirrhotic patients with ascites who require emergency room care or hospitalization, who demonstrate signs/symptoms suggesting SBP, or who present gastrointestinal bleeding, in order to exclude SBP. Several non-invasive methods were tried in many studies for SBP diagnosis, as alternatives to diagnostic paracentesis, e.g., fecal calprotectin. Moreover, numerous scores were proposed for SBP diagnosis with variable accuracies, such as procalcitonin, ESR, and CRP (PEC) index, the modified Wehmeyer SBP scoring system, and Mansoura scoring system. This study aims at evaluating the diagnostic accuracy of serum procalcitonin, PEC index, modified Wehmeyer, and Mansoura scoring systems for SBP in cirrhotic patients with ascites. participants will be subjected to: Clinical evaluation: medical history and physical examination, Routine Laboratory investigations, Serum procalcitonin, Ascitic fluid study, Ascitic fluid culture with antibiotic sensitivity, Abdominal ultrasonography. The following scores will be calculated: Modified Child Pugh score, MELD score, MELD Na score, PEC index, Modified Wehmeyer score, and Mansoura score.

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients with ascites

Exclusion Criteria:

Infections other than SBP.

* malignancy.
* Antibiotic therapy before hospital admission.
* Chemotherapy or radiotherapy within 1 month before admission.
* Pancreatic diseases.
* contraindication to paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Tropical Medicine and Gastroenterology Department
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
PEC index | five months
  procalcitoin × (ESR + CRP)
Modified Wehmeyer score | five months
  a score is calculated based on age, CRP level, and platelet count using a scale from 0 to 5 as follows: age >60 years: 1 point. platelet count <100,000/mL: 1 point CRP between 13.5 and30 mg/L: 1 point CRP between 30 and 60 mg/L: 2 points CRP above 60 mg/L: 3 points
Mansoura score | five months
  score is calculated based on age, mean platelets volume, neutrophil lymphocytic ratio, and CRP using a scale of 0 to 5 as follows: Age ≥55 years: 1 point MPV ≥8.5 fl: 1 point NLR≥2.5: 1 point CRP≥40 mg/l: 2 points

IPD SHARING:
Plan to Share IPD: No